CLINICAL TRIAL: NCT05478733
Title: Study of Factors Associated With Significant MYoCArdian Uptake on 68Ga-DOTATOC PET Scans for Oncology
Acronym: MYCADO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pierre Yves MARIE, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2021PI237
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Oncologic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chemotherapy-related cardiovascular morbidity and mortality in cancer patients is a public health concern. Although several imaging techniques exist to prevent and monitor chemo-induced cardiotoxic effects, the lack of recommendation and consensus is a barrier to reducing cardiac adverse events in this population. PET/CT with Gallium-68 somatostatin analogues (68Ga-DOTATOC, 68Ga-DOTATATE...) is now part of the reference imaging of neuroendocrine tumors (pulmonary, gastrointestinal, pancreatic, pheochromocytoma / paraganglioma, medullary thyroid cancer...), allowing to evaluate their extension and to follow up. Their treatment, including a large arsenal of chemotherapy (etoposide, capecitabine, cisplatin, etc.), may cause cardiotoxicity, which is difficult to assess.

DETAILED DESCRIPTION:
Chemotherapy-related cardiovascular morbidity and mortality in cancer patients is a public health concern. Although several imaging techniques exist to prevent and monitor chemo-induced cardiotoxic effects, the lack of recommendation and consensus is a barrier to reducing cardiac adverse events in this population. PET/CT with Gallium-68-labeled somatostatin analogues (68Ga-DOTATOC, 68Ga-DOTATATE...) is now part of the reference imaging of neuroendocrine tumors (pulmonary, gastrointestinal, pancreatic, pheochromocytoma/paraganglioma, medullary thyroid cancer...), allowing to evaluate their extension and to perform follow-up . Their treatment, including a large arsenal of chemotherapy (etoposide, capecitabine, cisplatin, etc.), may cause cardiotoxicity, which is difficult to assess. However, significant cardiac area uptake has been found on some 68Ga-DOTATOC PET/CT scans in oncology. This uptake could be related either to the patient's cardiac history (inflammatory atheromatous valvular and/or coronary lesions), some studies having shown the association between the uptake of a somatostatin analogue and the presence of calcified plaques, or to a possible chemo-induced cardiotoxicity which, to our knowledge, no study has investigated. Thus, the identification of 68Ga-DOTATOC binding patterns in the cardiac area in relation to chemo-induced cardiotoxicity would have the advantage of avoiding the multiplication of examinations in the initial and follow-up work-up, thus allowing the combined evaluation of the disease and the cardiac adverse effects induced by its treatments, and thus a better control of the cardio-induced morbidity and mortality of patients with a neuroendocrine tumor.

The hypothesis of this study is that 68Ga-DOTATOC PET/CT scans with oncological indications sometimes show significant uptake in the cardiac area, which could be related to inflammatory atheromatous coronary/valvular lesions, or to a recent history of potentially cardiotoxic oncological treatments (or to diffuse somatic inflammation?)

ELIGIBILITY:
Inclusion Criteria:

* patient having performed one or more 68Ga-DOTATOC PET/CT scans for oncology indications between 2019 and 2021 (23/01/2019 to 08/12/2021)
* patient who stayed in the nuclear medicine department between 2019 and 2021

Exclusion Criteria:

* patient with no oncological involvement

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient having performed one or more 68Ga-DOTATOC PET/CT scans for oncology indications
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Correlation between measurements and cardiac hyperfixation | 2 years
  Correlation between measurements of myocardial activity ratios and possible cardiac hyperfixation sites with blood activity and presence of cardiovascular history, and health data collected such as cardiovascular risk factors (and their number), and the existence of recent chemotherapy or radiotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: LAMBERT Aurélien, MD, MSc, Principal Investigator — ICL
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France